CLINICAL TRIAL: NCT04612413
Title: A Phase 2, Multi-Center, Randomized, Placebo-Controlled, Dose-Finding Study Evaluating Efficacy, Safety and Tolerability of Different Doses and Regimens of Allocetra-OTS for the Treatment of Organ Failure in Adult Sepsis Patients
Brief Title: A Phase 2 Study Evaluating Efficacy, Safety and Tolerability of Different Doses and Regimens of Allocetra-OTS for the Treatment of Organ Failure in Adult Sepsis Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Enlivex Therapeutics Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ENX-CL-02-002
Record Dates: First submitted 2020-10-26; First posted 2020-11-03 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Sepsis; Community-acquired Pneumonia; Urinary Tract Infections; Cholecystitis, Acute; Cholangitis Acute; Intraabdominal Infections
MeSH Terms: conditions — Sepsis; Community-Acquired Pneumonia; Urinary Tract Infections; Cholecystitis, Acute; Intraabdominal Infections

STUDY DESIGN:
Intervention Model Description: Up to Protocol Version 10.0, eligible patients were randomized to one of the 4 treatment groups in a 1:1:1:1 ratio between the 4 Cohorts:
  1. Placebo
  2. Single Intravenous (IV) dose of Allocetra-OTS, 5x10^9 cells
  3. Single IV dose of Allocetra-OTS, 10x10^9 cells
  4. Single or two IV doses of Allocetra-OTS, 10x10^9 cells in each dose
  Starting from Protocol Version 10.0, patient will be randomized to either Cohort 1 (Placebo) or Cohort 4 (Single or two IV doses of Allocetra-OTS, 10x10^9 cells in each dose).
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Cohort 1 (Placebo Comparator): Single IV dose of placebo solution
  Interventions: Other: Placebo
- Cohort 2 (Experimental): Single IV dose of 5x10^9 Allocetra-OTS cells in suspension
  Interventions: Drug: Allocetra-OTS
- Cohort 3 (Experimental): Single IV dose of 10x10^9 Allocetra-OTS cells in suspension
  Interventions: Drug: Allocetra-OTS
- Cohort 4 (Experimental): Single or two doses of 10x10^9 Allocetra-OTS cells in suspension
  Interventions: Drug: Allocetra-OTS

INTERVENTIONS:
Drug: Allocetra-OTS — Allocetra-OTS is a cell-based therapy consisting of non-HLA-matched allogeneic peripheral blood mononuclear cells, derived from a healthy human donor following a leukapheresis procedure, induced to an apoptotic stable state and suspended in a solution containing DMSO.
  Arms: Cohort 2; Cohort 3; Cohort 4
Other: Placebo — Solution containing all excipients except for the Allocetra-OTS cells
  Arms: Cohort 1

SUMMARY:
A Phase 2, Multi-Center, Randomized, Placebo-Controlled, Dose-Finding Study Evaluating Efficacy, Safety and Tolerability of Different Doses and Regimens of Allocetra-OTS for the Treatment of Organ Failure in Adult Sepsis Patients

DETAILED DESCRIPTION:
Allocetra-OTS is an immunomodulatory cell-based therapy consisting of allogeneic peripheral blood mononuclear cells that have been modified to be engulfed by macrophages and reprogram them into their homeostatic state.

This is a multi-center, randomized, placebo-controlled, dose-finding study comparing the efficacy, safety and tolerability of different dosing regimens of Allocetra-OTS, in patients with sepsis. The study aims to compare the safety and efficacy of different doses and regimens of Allocetra-OTS, as well as the clinical manifestations following Allocetra-OTS treatment, to that of Placebo in the treatment of organ failure in adult sepsis patients.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥18 years and ≤90 years of age.
2. Meets Sepsis 3 criteria with a SOFA score ≥5 above pre-admission status
3. Sepsis due to infection in at least one of the below organs:

   3.1. Community-Acquired Pneumonia (CAP). 3.2. Urinary tract infection 3.3. Acute cholecystitis diagnosed by Tokyo criteria 3.4. Acute cholangitis diagnosed by Tokyo criteria 3.5. Other intra-abdominal infections (IAI) 3.6. Skin or soft tissue infection
4. Adequate source control

Exclusion Criteria:

1. Sepsis due to infection other than lung infection, UTI, IAI, skin/soft tissue infection or sepsis patients where site of infection is unclear or unknown.
2. On chronic dialysis.
3. Patients with acute pancreatitis
4. Moribund patients
5. Weight <50 kg or >120 kg or BMI >40 kg/m^2.
6. SOFA score ≥14 at screening.
7. Patients with nosocomial infection.
8. A known malignancy.
9. Patients with end-stage disease (unrelated to sepsis)
10. Known active symptomatic SARS-CoV-2 or chronic viral infections, such as HBV or HCV, HIV or other chronic infections.
11. Chronic respiratory disease.
12. Known active upper GI tract ulceration or hepatic dysfunction.
13. Known NYHA class IV heart failure or unstable angina, ventricular arrhythmias, acute coronary disease or myocardial infarction.
14. Known immunocompromised state or medications known to be immunosuppressive.
15. Organ allograft or previous history of stem cell transplantation.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2020-11-30 (Actual); Primary Completion 2024-01-12 (Actual); Study Completion 2024-12-16 (Actual)

PRIMARY OUTCOMES:
Efficacy: Change from baseline in SOFA score | 28 days
  Change from baseline in SOFA score throughout 28 days
Safety: Number and severity of AEs and SAEs | 28 days
  Number and severity of AEs and SAEs throughout 28 days follow up period

SECONDARY OUTCOMES:
Ventilator-free days | 28 days
  Ventilator-free days over 28 days
Vasopressor-free days | 28 days
  Vasopressor-free days over 28 days.
Days without renal replacement therapy (dialysis). | 28 days
  Days without renal replacement therapy (dialysis).
Time in ICU and time in hospital | 28 days
  Time in ICU and time in hospital
Number of days with creatinine ≤ Baseline levels +20% | 28 days
  Number of days with creatinine ≤ Baseline levels +20%
All-cause mortality | 28 days
  All-cause mortality at Day 28 following first dose
Changes from baseline in CRP levels | 28 days
  Changes from baseline in CRP levels
Number and severity of AEs and Serious Adverse Events (SAEs) | 12 months
  Number and severity of AEs and Serious Adverse Events (SAEs) throughout 12 months follow up period
Detection of autoimmune and human leukocyte antigen (HLA) antibodies | 12 months
  Detection of autoimmune and human leukocyte antigen (HLA) antibodies

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Singer, MD, Principal Investigator — Rabin medical center, Belinson Campus, Petah Tiqwa Isarel
Locations (31):
- Belgium (4):
  - Clinique Saint-Pierre, Brussels
  - Saint-Luc Hospital University, Brussels
  - CHU de Charleroi, Charleroi
  - Ziekenhuis Oost-Limburg, Genk
- France (10):
  - CHU d'Angers, Angers
  - Vendee Departmental Hospital Center, La Roche-sur-Yon
  - University Hospital of Limoges, Limoges
  - CHU de Montpellier, Montpellier
  - CHU de Nantes, Nantes
  - Bretonneau Hospital, Paris
  - Centre Hospitalier Victor Dupouy, Paris
  - Reims University Hospital Robert Debre, Reims
  - CHU de Rennes, Rennes
  - Strasbourg University Hospital, Strasbourg
- Israel (7):
  - Soroka Medical Center, Beersheba
  - Hillel Yaffe Medical Center, Hadera
  - Bnai Zion Medical Center, Haifa
  - Hadassah Ein Kerem Medical Center, Jerusalem
  - Beilinson Medical Center, Petah Tikva
  - Ziv Medical Center, Safed
  - Poriya Medical Center, Tiberias
- Netherlands (2):
  - Canisius Wilhelmina Hospital, Nijmegen
  - Radboud UMC, Nijmegen
- Spain (8):
  - Clinic Barcelona University Hospital, Barcelona
  - University Hospital Sagrat Cor, Barcelona
  - Vall d'Hebron, Barcelona
  - Getafe University Hospital, Getafe
  - Dr. Josep Trueta University Hospital, Girona
  - University Hospital Arnau de Vilanova of Lleida, Lleida
  - General University Hospital Gregorio Maranon, Madrid
  - University Hospital Joan XXIII of Tarragona, Tarragona

IPD SHARING:
Plan to Share IPD: No